CLINICAL TRIAL: NCT07361627
Title: Improving Upper Limb Motor Control With Spinal Stimulation
Brief Title: Upper Limb Rehabilitation Using Non-invasive Spinal Cord Stimulation
Acronym: CIME_upperlimb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRIR 2024-2080
Record Dates: First submitted 2025-12-23; First posted 2026-01-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injury Cervical; Spinal Cord Injury, Acute; Spinal Cord Injury (Quadraplegia)
Keywords: Spinal cord injury; Sub-acute; Neuromodulation; transcutaneous Spinal Cord Stimulation; Activity-based therapy; Upper extremity motor score; Rehabilitation; Electroencephalography; EEG; Somatosensory evoked potential; Transcranial Magnetic Stimulation; Motor evoked potential; Clinical assessment; Neuroplasticity
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Intervention Model Description: The study model is a double-blind randomized controlled trial (RCT).
Who Masked: Participant, Outcomes Assessor
Masking Description: Clinical outcomes assessors and all participants are masked till the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity-based therapy with sham spinal stimulation (n=20) (Sham Comparator): Participants with cervical spinal cord injury (ASIA levels A-D) randomized to this arm will receive sham transcutaneous spinal cord stimulation combined with activity-based therapy. Training will consist of 20 sessions delivered over 6-8 weeks during the subacute stage.
  For the transcutaneous spinal cord stimulation (tSCS), a single or two self-adhesive cathode electrodes will be placed at the C4 to T1 vertebral levels. A pair of reference electrodes will be placed bilaterally on the external part of the clavicular regions. The stimulation will be set at minimal intensity, sufficient only for the participants to perceive it.
  Interventions: Other: Protocol 1: Combination of activity-based therapy and sham spinal cord stimulation
- Activity-based therapy with facilitatory spinal stimulation (n=20) (Experimental): Participants with cervical spinal cord injury (ASIA levels A-D) randomized to this arm will receive real-intensity transcutaneous spinal cord stimulation combined with activity-based therapy. Training will consist of 20 sessions delivered over 6-8 weeks during the subacute stage.
  For the transcutaneous spinal cord stimulation (tSCS), a single or two self-adhesive cathode electrodes will be placed at the C4 to T1 vertebral levels. A pair of reference electrodes will be placed bilaterally on the external part of the clavicular regions. The stimulation will be set at minimal intensity, sufficient only for the participants to perceive it. Individualized tSCS parameters (30-80Hz, 0-90mA, biphasic 400us pulse square) will be used to facilitate upper limb movement.
  Interventions: Other: Protocol 2: Combination of activity-based therapy and facilitatory transcutaneous spinal cord stimulation

INTERVENTIONS:
Other: Protocol 1: Combination of activity-based therapy and sham spinal cord stimulation — The training session for the sham group comprises of activity-based therapy along with sham stimulation on the spinal cord of the participants. These training sessions will include repetitive, intensive strength training and functional exercises targeting arm and hand (upper limb) movements. Sessions will be delivered by trained physiotherapists and occupational therapists. Each participant will complete 20 sessions over six to eight weeks (three per week), with each session lasting 45 minutes. Breaks will be added, if needed. Training will begin with a mental imagery exercise in which participants imagine performing a daily activity (e.g., drinking coffee in a café), followed by therapist-selected activities. Participants will receive transcutaneous spinal cord stimulation set at sensory threshold intensity (i.e., below the threshold that facilitates voluntary movement of the limb; usually 2-3 mA intensity), delivered simultaneously with training.
  Other Names: Sham stimulation
  Arms: Activity-based therapy with sham spinal stimulation (n=20)
Other: Protocol 2: Combination of activity-based therapy and facilitatory transcutaneous spinal cord stimulation — The training session for the experimental group comprises of activity-based therapy along with facilitatory stimulation on the spinal cord of the participants. These training sessions will include repetitive, intensive strength training and functional exercises targeting arm and hand (upper limb) movements. Sessions will be delivered by trained physiotherapists and occupational therapists. Each participant will complete 20 sessions over six to eight weeks (three per week), with each session lasting 45 minutes. Breaks will be added, if needed. Training will begin with a mental imagery exercise in which participants imagine performing a daily activity (e.g., drinking coffee in a café), followed by therapist-selected activities. Participants will receive transcutaneous spinal cord stimulation set at a target intensity that facilitates voluntary upper limb movement (usually between 10 and 25 mA) in the participants.
  Other Names: tSCS
  Arms: Activity-based therapy with facilitatory spinal stimulation (n=20)

SUMMARY:
The goal of this study is to evaluate if combining activity-based therapy (ABT) with transcutaneous spinal cord stimulation (tSCS) can improve recovery of arm and hand movement in people with cervical spinal cord injury (SCI). As secondary aims, the study will also investigate at how this combination approach affects the cortical changes in the somatosensory and motor areas of the brain, as well as in the spinal cord and whether it helps participants use their arms more in daily life.

The main questions relevant to this study are:

1. Is it feasible to use the ABT + tSCS combination for improving arm and hand movement more than ABT alone during the sub-acute stage after SCI?
2. Does ABT + tSCS induce neuroplasticity, that is, changes in the brain and spinal cord activity linked to motor and sensory functions?
3. Do participants who receive ABT + tSCS report greater use of their arms in daily activities compared to those who receive ABT only?

In this study, participants will:

* Receive either ABT + tSCS or ABT + sham stimulation (a low-intensity current that does not facilitate the movements)
* Take part in 20 training sessions over 6-8 weeks (3 times per week, 45 min of active training each). During this, they will perform strengthening, task-based training, and mental imagery exercises with a therapist.
* Complete clinical tests and neurophysiological assessments (transspinal electrical stimulation, electroencephalography and transcranial magnetic stimulation) at three time points-- at the start, after training, and one month later to measure recovery and brain activity changes.

Researchers will compare the assessment outcomes across the three time points.

DETAILED DESCRIPTION:
This study is led by Dorothy Barthélemy (Ph.D, pht, Principal Investigator (PI)), Marika Demers (Ph.D, erg., co-PI), Diana Zidarov (Ph.D, co-PI) and Sujata Sinha (PhD, postdoctoral fellow, project lead). Collaborator includes Victoria Duda (PhD).

Population: individuals with SCI with injury level above T2, falling into American Spinal Injury Association (ASIA) categories A to D, in the sub-acute phase, and of minimum age of 16 years. These participants are in-patients admitted in the Institut de réadaptation Gingras-Lindsay de Montréal, Canada.

Participants will be randomized (1:1 ratio) into two equal groups, ABT + tSCS and ABT + sham stimulation and stratified based on ASIA level, age and sex.

During the training session, the ABT + tSCS group will receive ABT combined with tSCS. The tSCS will be delivered using surface electrode placed between C4 and T1 as a cathode and self-adhesive surface electrodes placed in the clavicular region on both sides as anodes. tSCS will deliver tonic pulses (30 - 100 Hz) and at an intensity that facilitates voluntary movements (usually 15 mA and up), determined prior to the first training session. Each ABT session will include 5 parts:

1. Mental imaging exercises: participants will imagine the movement while following a sequence proposed by therapists.
2. Cardiovascular warm-up exercises: using equipment that will allow the participant to train their cardiovascular system.
3. Weight bearing and stretching exercises: exercises to prepare their upper body muscles for the strengthening exercises.
4. Muscle strengthening exercises: exercises to increase their strength, with adapted equipment if necessary.
5. Activity-based exercises: exercises composed of repetitive that are present in the participant's daily life.

In the ABT+ sham stimulation group, intensity will be set at sensory threshold that will not facilitate any movement (usually 2-3mA). The ABT will be similar to the other group.

Prior to the training, clinical tests will be conducted to assess assess their muscle strength, sensations, and the quality of movements participants can make with their arms. Specifically, the primary measure will consist of the Upper Extremity Motor Score from the with American Spinal Injury Association Impairment Exam. The secondary clinical measures will include the following assessments: the Grasp and Release Test, Monofilaments test, Sensory function of the upper limb dermatomes from C4 to T1, Grip and pinch strength with a dynamometer, Proprioception subtest of the Fugl Meyer Assessment, Tetraplegic Upper Limb Activity Questionnaire (TUAQ) and Finger-to-Nose Test from the Comprehensive Coordination Scale. More details of the measures are in the Outcome Measures section.

For neurophysiological measures, electrophysiological assessments will include transspinal evoked potential (TEP), motor evoked potentials (MEPs) using transcranial magnetic stimulation (TMS) and somatosensory evoked potentials (SSEPs) using electroencephalogram (EEG).

These assessments will be conducted before the training, immediately after the training and one month later.

As for the experiment, 40 participants will be recruited, as determined by a priori power analysis.

For the neuroplasticity evaluation, TEP, TMS and EEG will be used.

1. To assess the excitability of spinal pathways, the non-invasive procedure of single-pulse transcutaneous spinal stimulation (tSCS) will be used. Participants will be comfortably seated in a chair or in their wheelchair. Self-adhesive surface electrodes will be placed over the cervical spine, with the cathode (Dura stick plus double wire, Dura stick, USA) over C4-T1 and anodes over the external part of the clavicles (TENS electrodes, ROHVEMJ). Single-pulse tSCS will be delivered using a constant-current stimulator (DS8R, Digitimer, UK) to induce Transspinal evoked potentials (TEPs). Responses will be recorded from surface electromyography. More details of the measurement are in the Outcome Measures section.
2. To assess changes along the corticospinal tract (motor cortex projections to the spinal cord), a magnetic field using the TMS will be applied to the primary motor cortex (M1) over the representation area of the contralateral bicep brachii muscle (this is the target muscle). This response will be recorded painlessly using surface electromyography (EMG) electrodes placed over the targeted muscle. The entire evaluation, including setup, will take approximately one hour. The responses evoked by TMS, that is, the motor evoked potentials, (MEPs) will be compared across the 3 time frames in each group. Particularly, latency and peak-to-peak amplitude of MEPs will be measured. More details of the measurement are in the Outcome Measures section.

2. To assess changes in brain mechanisms, particularly those related to sensory function, EEG recordings will be performed using Brain Vision's 32-electrode cap, with the Fz electrode used as the reference. Recordings will be obtained using a Brain Vision 32-channel EEG cap referenced to Fz. The median nerve of the upper limb will be electrically stimulated to elicit cortical responses. The entire evaluation duration will be for 90 minutes including the setup.

EEG activity from C3 and C4 corresponding to the contralateral sensorimotor cortex, will be analyzed, focusing on the N20 and P25 somatosensory evoked potential (SSEP) components, which occur approximately 20 ms and 25 ms post-stimulus, respectively. The N20-P25 complex reflects transmission through ascending somatosensory pathways.

N20 refers to the SSEP peaking approximately 20 ms after the onset of electrical stimulation at the ulnar nerve. P25 follows the N20, peaking around 25 ms after stimulus onset. Together, these form the N20-P25 complex, which reflects the transmission along ascending neuronal pathways. The amplitude and latency of the SSEPs will be compared across the 3 time frames in each group. In addition to C3 and C4, the neighboring electrode regions will also be inspected to identify any additional SSEPs that may emerge. More details of the measurement are in the Outcome Measures section.

ELIGIBILITY:
Inclusion Criteria:

* quadraplegic participants with a subacute spinal cord injury (sSCI), defined as the stage of spinal cord damage occurring between 1 week and 6 months post-injury, that fall within the period of at least one year post-injury
* 16 years old or above
* have a lesion between above T2
* residual upper limb movement
* have injury level according to ASIA A to D
* hospitalized in the hospital linked with the research center at Gingras Lindsay Rehabilitation Institute of Montreal, 6300 Darlington, Montreal
* can provide informed consent (no severe cognitive deficits by MoCA)
* be able to follow instructions in French or English

Exclusion Criteria:

* have a pacemaker
* have active cancer on stimulation site or metastatic cancer
* have unstable health conditions
* have unhealed wound, scar or pain which makes positioning of the electrodes impossible
* participants with specific contraindications to TMS (epilepsy, non-union cranial fracture and increased intracranial pressure) will be able to participate in the study, but will not receive TMS

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-08-09 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Motor Score (UEMS) | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  This will be used for assessing the motor function, that is, the strength and functionality of the muscles involved in movement. It helps determine the severity of motor impairments in patients with cervical lesions and is used to track recovery and assess outcome during inpatient rehabilitation. It has high inter-rater and intra-rater reliability. It also has high validity as an impairment measure and has moderate validity for predicting real-world functional independence.
  The test evaluates five movements of each arm, namely, elbow flexion, wrist extension, elbow extension, middle finger flexion, and little finger abduction. The participant is asked to perform these movements either actively or passively, depending on their ability. These are scored on a scale from 0 (no movement) to 5 (full function). Thus, the higher score reflects improvement in the motor function across the three time frames.

SECONDARY OUTCOMES:
Grasp and Release Test | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  This will be used to assess hand motor skills and the ability to pick up, move and release 6 objects of different sizes, weights and textures. This includes lateral prehension for peg, paperweight and fork, and palmar prehension for block, can and videotape.
  The test has high inter-reliability and test-retest reliability for each object and a strong intra-rater reliability. It also has a good construct validity (scores correlate with motor strength and hand function), high convergent validity with activities of daily living test, and moderate to high predictive validity.
  Participants must use their hand without prosthesis to grasp an object and release it in a box (rotation of limb is not permitted). This is repeated several times, and the number of successful grasp-release is recorded. Sequence is completed as many times as possible during 30 seconds, for each object (3-5 trials per object) with 30 seconds rest between two objects.
Dermatome (sensory) test | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  This will be used to assess the sensory level of the participant by evaluating the ability to feel stimuli and to differentiate between sharp and dull sensations (pinprick test) on specific regions of the skin corresponding to spinal nerve segments.
  The summed sensory scores (light touch + pinprick) have good to excellent inter- and intra-rater reliability. So, we will use the summed scores. The test has good validity for classifying lesion level and severity, moderate for predicting function, and has limited sensitivity (not sensitive to subtle changes) compared to electrophysiological or quantitative tests.
  Light touch and pinprick sensation are first demonstrated on the participant's cheek. The participant, seated with eyes closed, is tested using light touch with tissue or cotton (assessing large A fibers) and pinprick with a pin or toothpick (assessing smaller A-delta and C fibers for superficial pain) at six test sites. The sensation is reported by them.
Monofilament test | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  This will be used to quantify and to assess the sensory function, particularly for detecting areas of sensory loss or abnormal sensation (neuropathic pain). This test has high validity and inter-and intra tester reliability in participants with chronic cervical spinal cord injury.
  The test is conducted using Semmes-Weinstein monofilaments. With eyes closed, the participant is asked to report whether they can feel the pressure when a monofilament is applied to different regions of the upper limb. The threshold at which the stimulus is perceived is recorded (5.88, 5.07, 4.56, 4.08, 3.22). Specific regions are assessed depending on the nerve: the pulp of the middle finger for the median nerve, the pulp of the little finger for the ulnar nerve, the first dorsal space of the hand between the thumb and index finger and the lateral epicondyle at the extensor compartment for the radial nerve, and the deltoid region for the axillary nerve.
Force (Grip and Pinch Strength) test | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  This will be used to assess grip and pinch strength which are used in daily tasks involving hand function. The Pinch strength test has good to excellent reliability for neurological conditions and has strong to very strong correlations with grip strength. It has a good validity.
  The Grip strength has an excellent test-retest reliability in SCI. It shows a very high intra- and inter-rater reliability if standardized protocols (same dynamometer, position, instructions) are followed. It has a good validity.
  Grip strength is measured using a dynamometer, with the participant seated and the elbow flexed at 90 degrees. The participant must squeeze the device as hard as possible for 3 trials; the average of these trials is calculated. Pinch strength is measured using a pinch gauge, where the participant pinches an object between the thumb and index finger with maximum effort. Again, the average of 3 trials is taken.
Proprioception | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  This test is used to the assess the ability to sense the position of the limbs in space, important for evaluating proprioceptive deficits that can affect balance and coordination.
  It has a moderate overall and inter-rater reliability and depends strongly on the therapist's technique. Intra-rater reliability is better but is variable as participants can have fatigue or guess. Test-retest reliability is lower than that of dermatomes or motor scores.
  It has a limited validity; construct validity is supported and concurrent validity shows moderate correlation with function; criterion validity is limited.
  The participant is blinded while the therapist moves their upper limb (shoulder, elbow, and wrist) to a specific position and asks them to replicate the position with the opposite limb or to report the position. Results are reported as the difference between the actual and replicated positions.
Coordination test | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  This test is used to assess the ability to perform smooth, controlled movements, critical for fine motor tasks (e.g. writing, buttoning a shirt).
  Its reliability is generally low to moderate: intra-rater reliability is variable as it depends on the therapist scoring, inter-rater reliability is moderate at best, and test-retest reliability is limited since coordination can fluctuate with fatigue, spasticity, or attention.
  Validity is also limited, with moderate construct validity, low to moderate concurrent validity, and limited criterion validity.
  The standard finger-to-nose test is used: the participant is asked to touch a target with the index finger and then their nose, repeating the movement five times at a fast but comfortable pace. The therapist observes for tremors, uncoordinated movements, delays, and scores performance using a 12-point scale per side that considers precision, fluidity, arm movement, and trunk stability.
Transspinal evoked potentials (TEPs) | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  TEPs will be measured through single-pulse transcutaneous spinal stimulation (tSCS). The cathode (Dura stick plus double wire, Dura stick, USA) will be positioned at the midline over C4-T1 and anode over the external part of the clavicles (TENS electrodes, ROHVEMJ). Single-pulse tSCS will be delivered using a constant-current stimulator (DS8R, Digitimer, UK) with monophasic square-wave pulses of 1ms at a frequency of 0.2Hz to induce TEPs. Responses will be recorded from surface electromyography. Stimulation intensity will be gradually increased from 0 to evoke a potential in all, or in the maximum number of upper limb muscles recorded. Two of the outcome measures will be for each muscle: the motor threshold, i.e., the lowest intensity inducing 5/10 stimulation responses; and the recruitment curve. The third measure will include amplitude, latency, and duration of the TEP at 120% of the motor threshold, determined for the myotome that showed the smallest response.
Transcranial magnetic stimulation (TMS)- motor evoked potentials | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  This neurophysiological assessment will be done to test if there are neuroplastic changes because of the ABT + tSCS training. TMS will be applied to the primary motor cortex (M1) over the representation area of the contralateral bicep brachii muscle (this is the target muscle). A figure-8 shaped coil will deliver the magnetic field to activate motor nerves, leading to the activation of the target muscle. This response will be recorded painlessly using surface electromyography electrodes placed over the targeted muscle. Four 5-minute stimulation sets, each separated by 2-minute rest periods, will be conducted. The entire evaluation, including setup, will take approximately one hour. The responses evoked by TMS, that is, the motor evoked potentials, (MEPs) will be compared across the 3 time frames in each group. Quantitative parameters will include MEP amplitude (magnitude), and latency, serving as indicators of cortico-spinal excitability changes pre- and post-intervention.
Electrophysiology (EEG)-Somatosensory evoked potentials (SSEPs) | 3 time points: Pre-intervention (Day 0, prior to the first training session), Post-intervention (+/-1 week) and one-month post-intervention (+/- 1 week).
  This test will also be done for neuroplastic evaluation. SSEPs are time-locked EEG responses reflecting sensory pathway conduction from peripheral nerves to the somatosensory cortex. Participants will be comfortably seated in a chair. For each arm, the median nerve will be stimulated using surface electrodes placed near the wrist to elicit upper-limb SSEPs. EEG will be recorded with a 32-channel cap (Brain Vision Recorder 2.0) following the 10-20 system, referenced to Fz. During a 10-minute session for each arm, 1800 stimuli (3 Hz, 0.001 s duration) will be delivered at 5% of the maximal flexor carpi radialis response. EEG signals will be sampled at 5000 Hz and analyzed in BrainVision Analyzer using filtering and averaging. Primary regions of interest include C3/C4 and adjacent electrodes (Cz, C1/2, FCz). The expected SSEPs are N20 (~20 ms) and P25 (~25 ms). The presence, amplitude, and latency of the N20-P25 complex will serve as measures of somatosensory pathway excitability.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Barthelemy, pht., PhD, Principal Investigator — Université de Montréal
Locations (1):
- Institut de réadaptation Gingras-Lindsay-de-Montréal (IRGLM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynskey JV, Belanger A, Jung R. Activity-dependent plasticity in spinal cord injury. J Rehabil Res Dev. 2008;45(2):229-40. doi: 10.1682/jrrd.2007.03.0047. PMID 18566941
- [Background] Steele AG, Manson GA, Horner PJ, Sayenko DG, Contreras-Vidal JL. Effects of transcutaneous spinal stimulation on spatiotemporal cortical activation patterns: a proof-of-concept EEG study. J Neural Eng. 2022 Jul 1;19(4). doi: 10.1088/1741-2552/ac7b4b. PMID 35732141
- [Background] Manson G, Atkinson DA, Shi Z, Sheynin J, Karmonik C, Markley RL, Sayenko DG. Transcutaneous spinal stimulation alters cortical and subcortical activation patterns during mimicked-standing: A proof-of-concept fMRI study. Neuroimage Rep. 2022 Jun;2(2):100090. doi: 10.1016/j.ynirp.2022.100090. Epub 2022 Mar 8. PMID 36212800
- [Background] Dimitrijevic MR, Illis LS, Nakajima K, Sharkey PC, Sherwood AM. Spinal cord stimulation for the control of spasticity in patients with chronic spinal cord injury: II. Neurophysiologic observations. Cent Nerv Syst Trauma. 1986 Spring;3(2):145-52. doi: 10.1089/cns.1986.3.145. PMID 3490313
- [Background] Sadowsky CL, McDonald JW. Activity-based restorative therapies: concepts and applications in spinal cord injury-related neurorehabilitation. Dev Disabil Res Rev. 2009;15(2):112-6. doi: 10.1002/ddrr.61. PMID 19489091
- [Background] Murray LM, Knikou M. Transspinal stimulation increases motoneuron output of multiple segments in human spinal cord injury. PLoS One. 2019 Mar 7;14(3):e0213696. doi: 10.1371/journal.pone.0213696. eCollection 2019. PMID 30845251
- [Background] Kalsi-Ryan S, Beaton D, Curt A, Popovic MR, Verrier MC, Fehlings MG. Outcome of the upper limb in cervical spinal cord injury: Profiles of recovery and insights for clinical studies. J Spinal Cord Med. 2014 Sep;37(5):503-10. doi: 10.1179/2045772314Y.0000000252. PMID 25229734
- [Background] Wuolle KS, Van Doren CL, Thrope GB, Keith MW, Peckham PH. Development of a quantitative hand grasp and release test for patients with tetraplegia using a hand neuroprosthesis. J Hand Surg Am. 1994 Mar;19(2):209-18. doi: 10.1016/0363-5023(94)90008-6. PMID 8201183
- [Background] Velstra IM, Bolliger M, Baumberger M, Rietman JS, Curt A. Epicritic sensation in cervical spinal cord injury: diagnostic gains beyond testing light touch. J Neurotrauma. 2013 Aug 1;30(15):1342-8. doi: 10.1089/neu.2012.2828. PMID 23895137
- [Background] Sullivan KJ, Tilson JK, Cen SY, Rose DK, Hershberg J, Correa A, Gallichio J, McLeod M, Moore C, Wu SS, Duncan PW. Fugl-Meyer assessment of sensorimotor function after stroke: standardized training procedure for clinical practice and clinical trials. Stroke. 2011 Feb;42(2):427-32. doi: 10.1161/STROKEAHA.110.592766. Epub 2010 Dec 16. PMID 21164120
- [Background] Molad R, Alouche SR, Demers M, Levin MF. Development of a Comprehensive Outcome Measure for Motor Coordination, Step 2: Reliability and Construct Validity in Chronic Stroke Patients. Neurorehabil Neural Repair. 2021 Feb;35(2):194-203. doi: 10.1177/1545968320981943. PMID 33410389
- [Background] Tefertiller C, Rozwod M, VandeGriend E, Bartelt P, Sevigny M, Smith AC. Transcutaneous Electrical Spinal Cord Stimulation to Promote Recovery in Chronic Spinal Cord Injury. Front Rehabil Sci. 2021;2:740307. doi: 10.3389/fresc.2021.740307. Epub 2022 Jan 4. PMID 36004322
- [Background] Gopaul U, Bayley MT, Kalsi-Ryan S. Combined Activity-Based Therapy and Cervical Spinal Cord Stimulation: Active Ingredients, Targets and Mechanisms of Actions to Optimize Neurorestoration of Upper Limb Function After Cervical Spinal Cord Injury. Physiother Res Int. 2025 Apr;30(2):e70036. doi: 10.1002/pri.70036. PMID 39927575
- [Background] Mulcahey MJ, Betz RR, Kozin SH, Smith BT, Hutchinson D, Lutz C. Implantation of the Freehand System during initial rehabilitation using minimally invasive techniques. Spinal Cord. 2004 Mar;42(3):146-55. doi: 10.1038/sj.sc.3101573. PMID 15001979
- [Background] Marino RJ, Jones L, Kirshblum S, Tal J, Dasgupta A. Reliability and repeatability of the motor and sensory examination of the international standards for neurological classification of spinal cord injury. J Spinal Cord Med. 2008;31(2):166-70. doi: 10.1080/10790268.2008.11760707. PMID 18581663